CLINICAL TRIAL: NCT05474586
Title: A Randomised, Double-blind, Placebo-controlled Study to Evaluate the Efficacy and Safety of Collavant n2 in Individuals With Osteoarthritis of the Knee
Brief Title: To Evaluate the Efficacy and Safety of Collavant n2 in Individuals With Osteoarthritis of the Knee
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Vedic Lifesciences Pvt. Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: BI/210903/COLL/OA
Record Dates: First submitted 2022-07-22; First posted 2022-07-26 (Actual); Last update posted 2023-09-06 (Actual); Status verified 2023-09

CONDITIONS: Osteoarthritis, Knee
MeSH Terms: conditions — Osteoarthritis, Knee | interventions — Glucosamine; Chondroitin Sulfates; microcrystalline cellulose

STUDY DESIGN:
Intervention Model Description: Randomized, Parallel Group, Placebo Controlled Trial
Who Masked: Participant, Care Provider, Investigator
Masking Description: Sequentially numbered, sealed, opaque envelopes
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Collavant n2 40 mg/day (Experimental): 2 capsules in the morning before breakfast and 2 capsules at night before going to bed for 180 days
  Interventions: Other: Collavant n2 40 mg/day
- Glucosamine hydrochloride & Chondroitin sulfate (Active Comparator): 2 capsules in the morning before breakfast and 2 capsules at night before going to bed for 180 days
  Interventions: Other: Glucosamine hydrochloride & Chondroitin sulfate
- Microcrystalline cellulose (Placebo Comparator): 2 capsules in the morning before breakfast and 2 capsules at night before going to bed for 180 days
  Interventions: Other: Microcrystalline cellulose

INTERVENTIONS:
Other: Collavant n2 40 mg/day — 2 capsules in the morning before breakfast and 2 capsules at night before going to bed for 180 days
  Arms: Collavant n2 40 mg/day
Other: Glucosamine hydrochloride & Chondroitin sulfate — 2 capsules in the morning before breakfast and 2 capsules at night before going to bed for 180 days
  Arms: Glucosamine hydrochloride & Chondroitin sulfate
Other: Microcrystalline cellulose — 2 capsules in the morning before breakfast and 2 capsules at night before going to bed for 180 days
  Arms: Microcrystalline cellulose

SUMMARY:
A randomised, double-blind, placebo-controlled study to evaluate the efficacy and safety of Collavant n2 in individuals with osteoarthritis of the knee.

ELIGIBILITY:
Inclusion Criteria:

1. Male and females ≥ 40 to ≤ 75 years suffering from knee joint pain for atleast 3 months before screening.
2. Body mass index (BMI) ≥ 18.5 and ≤ 29.9 kg/m2
3. Pain VAS for knee joint pain ≥ 5 and ≤ 7 cm on a 10 cm scale at screening.
4. Radiographic evidence of grade II/III knee OA based on the Kellgren and Lawrence (KL) radiographic entry criteria for OA - i Grade II: Antero-posterior weight-bearing knee radiograph demonstrates possible joint space narrowing (JSN) with definite osteophyte formation.

   ii Grade III: Antero-posterior weight-bearing knee radiograph demonstrates definite joint space narrowing, multiple osteophyte formations, some sclerosis, and possible deformity of bony ends.
5. LAI score of ≥ 6 - ≤10 at screening.
6. Willing to stop the restricted dietary supplements, home-based remedies, and any other form of topical products or medications for knee joint pain relief or any other reason for the entire study duration.

   (Note: only hot and cold fomentation will be allowed, and the participant has to record the daily frequency of fomentation in the diary. The hot/cold fomentation needs to be stopped 48 hours prior to all assessment visits.)
7. Willing to stop using rescue medication 48 hours prior to all assessment visits.
8. Using the western toilet at home and/or workplace.
9. Willingness to participate and comply with the study procedures and required visits.
10. Ability to understand and sign a written informed consent form, which must be completed before performing study-specific tasks.
11. Literate and have the ability to complete the study-based questionnaires and tasks.
12. Female participants of childbearing age must be willing to use the acceptable methods of contraception during the study.

Exclusion Criteria:

1 History of uncontrolled hypertension and/or systolic blood pressure ≥ 140 mmHg and/or diastolic blood pressure ≥ 90 mmHg. 2 Fasting blood glucose (FBG) > 125 mg/dl. 3 Radiographic evidence of Grade I or Grade IV OA based on the KL radiographic criteria for osteoarthritis. 4 Any history of trauma, fractures, or surgery to the index joint. 5 Any planned surgery (diagnostic or therapeutic intervention) to the index joint during the participation in the study. 6 History of use of corticosteroid, disease modifying drugs, glucosamine, chondroitin, and intra-articular treatments including injections of corticosteroid or hyaluronic acid within 6 months of the screening visit and consumption of Omega-3 fatty acids or other joint health supplements within 15 days preceding the screening visit. 7 History of use of gabapentin within 6 weeks and/or methylcobalamin within 2 weeks prior to screening. 8 Known case of deformity of the knee joint or diagnosed on clinical examination during screening. 9 Known case of any joint disorder involving the index joint that includes but is not limited to known rheumatic or inflammatory conditions such as rheumatoid arthritis, osteomyelitis, osteoporosis, severe OA, and bone metastasis. 10 Known cases of gout and/or hyperuricemia (serum uric acid >440 μmol/L). 11 Other pathologic lesions on X-ray of the knee. 12 History of bleeding disorders (e.g., Haemophilia, Sickle cell anaemia, etc.).

13 Participants with abnormal levels of serum thyroid-stimulating hormone (TSH) (< 0.4 to > 4.2 mIU/L). 14 Any history or evidence of allergy to chicken, eggs, or protein products in the past. 15 Alcoholics or known drug dependents. (Alcoholism or heavy alcohol use is interpreted based on alcohol content consumed per day or week. It is defined as more than 4 drinks on any day or more than 14 drinks per week for men. For women, it is defined as more than 3 drinks on any day or more than 7 drinks per week. Standard alcoholic drink is roughly equivalent to 14 grams of pure alcohol, which is found in the following: i 12 ounces (Approx. 350 ml) of regular beer, which is usually about 5% alcohol ii 5 ounces (Approx. 150 ml) of wine, which is typically about 12% alcohol iii 1.5 ounces (Approx. 45 ml) of distilled spirits, which is about 40% alcohol) 16 History of smoking or currently smoking or using any form of smokeless tobacco. 17 Not willing to abstain from the use of NSAIDs (including low dose aspirin 50 mg/day for cardiovascular health). 18 Participation in a study of an investigational product within 90 days prior to the screening.

Ages: 40 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 236 (Actual)
Dates: Start 2022-08-08 (Actual); Primary Completion 2023-07-04 (Actual); Study Completion 2023-07-04 (Actual)

PRIMARY OUTCOMES:
Western Ontario and McMaster Universities Osteoarthritis Index Pain subscale | Day 0, 7, 30, 60, 90, 120, 150, and 180
  Knee joint pain as assessed by the change in the Western Ontario and McMaster Universities Osteoarthritis Index Pain subscale (WOMAC-P) score.
  the primary efficacy variable for the present study is the total WOMAC index score, the scores for each subscale will be summed up (Pain range: 0-20, Stiffness range: 0-8, and Physical function range: 0-68). Thus, the total WOMAC score will range from 0 - 96.
  The lowest the score is the good response and highest the score is extreme pain i.e. bad response.

SECONDARY OUTCOMES:
Knee joint pain as assessed by the change in the Western Ontario and McMaster - Pain subscale score. | Day 0, 7, 30, 60, 90, 120, 150, and 180
  The first domain, WOMAC-P, comprises 5 questions evaluating the amount of pain due to OA in the index joint experienced by the participant. The WOMAC-P subscale score of 0 indicates 'No pain' and 4 indicates 'Extreme pain'.
Knee joint stiffness as assessed by the change in the WOMAC - Stiffness subscale (WOMAC-S) score. | Day 0, 7, 30, 60, 90, 120, 150, and 180
  The domain, WOMAC-S, consists of 2 questions evaluating the amount of stiffness (resistance of the joint to movement characterized by difficulty in moving the joint along with pain and discomfort in the joint) experienced in the index joint. On the Likert scale, 0 indicates 'No stiffness' and 4 indicates 'Extreme stiffness'.
Knee joint function as assessed by the change in the WOMAC - Physical function (WOMAC-PF) score. | Day 0, 7, 30, 60, 90, 120, 150, and 180
  The WOMAC-PF consists of 17 questions evaluating the degree of physical difficulty experienced in the index joint due to OA in the third domain. For WOMAC-PF, 0 indicates 'No difficulty' and 4 indicates 'Extreme difficulty'.
Knee joint pain assessed by the change in the Visual Analogue Scale (VAS) score. | Day 0, 7, 30, 60, 90, 120, 150, and 180
  Point 0 indicates no pain and 10 indicates worst pain.
Severity of osteoarthritis as assessed by the change in the Lequesne algofunctional index (LAI) score. | Day 0, 7, 30, 60, 90, 120, 150, and 180
  Higher scores indicate a worse joint condition and Lowest scores indicate agood joint condition

CONTACTS AND LOCATIONS:
Overall Officials: Dr Shalini Srivastava, MD medicine, Study Director — Vedic Lifesciences Pvt. Ltd.
Locations (10):
- India (10):
  - Amber Clinic, Ahmedabad, Gujarat
  - Prme Orthopedic Speciality, Mumbai, Maharashtra
  - Diamond Hospital, Mumbai, Maharashtra
  - Ayush Nursing Home, Mumbai, Maharashtra
  - Life Care Hospital, Nashik, Maharashtra
  - Sparsh Hospital, Panvel, Maharashtra
  - Care n Cure Multispeciality Hospital, Pālghar, Maharashtra
  - Lifepoint Multispeciality Hospital, Pune, Maharashtra
  - Imperial Multispecialty Hospital, Pune, Maharashtra
  - Gayatri Hospital, Vasai, Maharashtra

IPD SHARING:
Plan to Share IPD: Undecided